CLINICAL TRIAL: NCT05259059
Title: Feeding Mom Feeding Infant's Microbiota: Nutritional Strategies for Improving Breast Milk Composition and Infant Health
Status: Recruiting | Type: Observational
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, Prof. WONG Man Sau, Professor, The Hong Kong Polytechnic University
Other Study IDs: HSEARS20211018004
Record Dates: First submitted 2022-02-07; First posted 2022-02-28 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: Breastfeeding; Infant Development
Keywords: Early nutrition; Breastfeeding; Infant growth
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — During the interviews at 3rd and 6th month postpartum, each breastfeeding mother will supply a specimen of breast milk in a private interview room. Peripheral venous blood will be collected from mothers at 3rd or 6th month postpartum. Infant urine and feces will be collected on diapers at 3rd, 6th and 12th month visit.
  Genes that relates to breastmilk secretion including Fucosyltransferase 2 and Fucosyltransferase 3, as well as 16S ribosomal deoxyribonucleic acid sequencing of the infant fecal samples would be determined analyzed from the collected sample.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention is involved — No intervention is involved

SUMMARY:
The first 1000 days, i.e., the earliest stage of life, is a unique period of opportunity to establish the foundations of human growth and health through the lifespan. In the recent decades, multiple studies have explored nutritional strategies for improving infant health through improving the nutritive and bioactive compositions in breast milk. For example, dietary fiber intake has been increasingly reported to benefit the health of the mother-infant dyad. However, the complex interplays among maternal diet, breast milk composition, infant gut microbiota and infant development are yet to be elucidated in a prospective cohort. In addition, the investigators' previous work has revealed unsatisfactory dietary patterns in Hong Kong lactating women, with clear inadequacy in fruit and vegetable intake. In this prospective cohort study, the investigators aim to recruit 100 healthy Chinese mother-child pairs. Data on maternal and infant dietary intake, breast milk composition, gut microbiota profile will be collected and the investigators will examine their associations with the health outcomes in infants. In addition, the influence of dietary factors and genetic predisposition on breast milk components and its associated benefits in the child will be interrogated. With the employment of multidisciplinary research approaches, cutting-edge biotechnologies and the omics platforms, this project will provide novel insights into the dietary factors and breastfeeding practices that are beneficial to the infant developmental trajectory, and the potential roles of breast milk composition in shaping infant's gut microbiota and the associated health impact in the long term. More importantly, the investigators hope to generate more solid scientific data to inform the public of the importance of maternal diet and the practical nutritional strategies to improve breast milk composition for the sake of the child.

DETAILED DESCRIPTION:
The First 1,000 Days approach highlights the time between conception and a child's second birthday as a critical period where adequate nutrition is essential for adequate development and growth throughout the child's life and potentially onto their own offspring. Childhood and adulthood health risks may be primed by nutritional status during this period.

In recent decades, accumulating evidence shows that gut microbiota plays indispensable roles in programming the growth, immunity and metabolic capacity of a person since birth. In addition, gut microbiota also exerts a significant impact on the disease risks at a later life stage, e.g., the development of obesity and cardiometabolic disorders. As such, factors (e.g., breast milk composition, exposure to antibiotics) that influence the initial establishment of gut microbiome during infancy and childhood should be carefully considered and optimized. It has now been determined that breast milk, as the sole nutrient source for infant, has a major impact in shaping early gut microbiota. However, there is still limited understanding on the complex interplay among maternal diet, feeding practices and infant health outcomes including the gut microbiota which are keys to the infant's developmental trajectory.

Maintaining a balanced diet with varieties of food is important to both the lactating mother and her child. In addition to rich nourishment from animal-based foods, plant-based diet provides an additional wide array of nutrients and bioactive components. First, dietary fiber, abundant in multiple plant-based foods, is beneficial to metabolic health, strengthening oxidative defense and profile of blood glucose, insulin sensitivity and blood lipid. Through the fermentation of gut microbiota in distal intestine, dietary fiber can be converted into multiple types of short chain fatty acids (SCFAs), which are involved in multiple physiological functions, and may enhance gut microbiota diversity and functionality. Second, as many bioactive phytochemicals are bound to macromolecules such as polysaccharides, fiber-rich foods are also good sources of phyto-nutrients including polyphenols and carotenoids. As well referenced before, flavonoids and carotenoids are established biomarkers for the intake of fruits and vegetables whose metabolites can be found in urine and breast milk. In the investigators' pilot analysis among nine lactating women, the investigators have found a significant inverse correlation between fiber intake during late trimester and infants' stool microbiota abundance of Firmicutes at 2nd month postpartum, the phylum of bacteria which might relate to a lower risk of cardiometabolic diseases. However, how maternal intake of plant-based foods affects the production and composition of breast milk in lactating women and the infant's gut microbiome is yet to be clarified.

Through increasing the intake of plant-based foods for lactating women, it may also provide micronutrients that are important for infants. For instance, omega-3 fatty acids and vitamin A are essential nutrients for infants' visual development. Flaxseed oils, walnuts and chia seeds are the common plant-based sources of alpha-linoleic acid, the precursor of eicosapentaenoic acid (EPA) and docosahexaenoic acid (DHA). DHA is highly concentrated in the photoreceptor outer segment membranes of the retina, and is essential for visual function. Apart from omega-3 fatty acids, vitamin A involves in visual transduction and the formation of visual pigments. Vitamin A is a group of organic compounds that includes retinol, retinal, and several provitamin A (carotenoids), which can be commonly found in orange and yellow vegetables and fruits (e.g. carrots, peaches, corns), and most dark green, leafy vegetables. Several carotenoids (beta-carotene, lutein, ß-cryptoxanthin and zeaxanthin) may reduce the long-term risk of cataract.

Despite the important role of maternal nutrition during pregnancy and breastfeeding periods and the long-term health of both mother and the offspring, there has been limited data in Hong Kong. In the investigators' pilot study among 64 mother-child pairs, the investigators examined the maternal diet in late pregnancy and found that only 10.0% and 25.0% of participating mothers have met the dietary recommendation on dietary fiber (25 grams/day) and vitamin A (770 μg of retinol activity equivalents/day) intake. Although the results might not fully represent the Hong Kong population, the inadequate intake of dietary fiber from plant-based foods for Hong Kong mothers warrants concern.

In the recent years, the Hong Kong society has increasing awareness on the importance of breastfeeding, and the initiation rate for breastfeeding was 87.5% in 2018. The improved rate of breastfeeding has been attributed by the collaborative efforts from various healthcare professionals, including physicians, nurses and lactating consultants, through the delivery of training sessions and frequent follow-up. However, the focus in current practice in clinical setting is to initiate and maintain breastfeeding practice, but fewer attention has been paid to optimize the nutrient composition in breast milk. Given that vitamin A is transferred to offspring by limited placental transfer during gestation, and mostly through breast milk during lactation, inadequate maternal intake of vitamin A and/or provitamin A may put infants at risk of deficiency. In another pilot study, the investigators have compared retinol and selected carotenoid contents in breast milk from 92 Hong Kong lactating mothers with high (3.0 servings/day on average) or low (1.2 servings/day on average) vegetable intakes, and mothers that consumed ß-carotene-containing supplements (2.4 servings of vegetables/day on average). The results showed that supplement users had significantly higher ß-carotene and retinol levels in breast milk, while mothers with higher vegetable intakes had significantly higher lutein levels in breast milk, and vegetable intake significantly correlated with the availability of lutein, ß-carotene, and lycopene in breast milk. Taken together, improving maternal diet may provide better nutrient composition in breast milk, and prevent low nutritional status of mothers.

In brief, many previous studies on the relationship between maternal diet, bioactive components in breast milk and infant health outcomes were cross-sectional in nature, while the inter-relationships between maternal diet, breast milk composition, infant gut microbiota and infant development warrants further clarification. How maternal dietary factors and infant feeding practices during the early life may influence the health outcomes infants is another perspective that worth examination. From the perspective of nutritional epidemiology, a high-quality prospective cohort will be needed to provide strong evidence to verify food-based dietary practices for postpartum women (e.g., the consumption of whole-grain cereals, fruits, and vegetables as recommended by the World Health Organization Global Strategy on Diet, Physical Activity, and Health) that may improve the general health of mothers and their children. Therefore, the investigators proposed a prospective cohort to uncover the underlying linkage among maternal diet, breast milk composition, gut microbiota and infant developmental conditions through a multi-omics approach.

ELIGIBILITY:
Inclusion Criteria for Mothers:

1. Hong Kong residents aged 18-40 years old;
2. Vaginal delivery between 37 and 42 weeks of gestation;
3. Carrying a singleton pregnancy;
4. Breastfeeding for >80% feeding occasions upon recruitment;
5. Intend to continue breastfeeding at least till the infant reaches 3-month old;

Inclusion Criteria for Infants:

1. Delivered between 37 and 42 weeks;
2. Born by vaginal delivery;
3. Singleton infant with no known abnormality;

Exclusion Criteria:

1. Complicated pregnancy such as preeclampsia and gestational diabetes;
2. Special dietary restrictions for examples gluten-free diets, vegan or any restrictions due to food allergies;
3. Suffer from renal, liver, or thyroid dysfunction, cognitive impairment, or any other indication of a major medical or psychological illness, as judged by the investigators as ineligible to participate the study
4. Have no intention to continue breastfeeding beyond 3 months.

Ages: 1 Month to 40 Years | Sex: All
Age Groups: Child, Adult
Gender Based: Yes — the subjects are mothers and their infants so female subjects needed to be selected while there is no sex limitation in the infants
Study Population: They are Hong Kong lactating women and their infants. Both of them are healthy and intend to continue breastfeeding at least 3 months.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-04-19 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
The consumption of dietary fiber in grams by participants | through study completion, an average of 1 year
  Dietary fiber intake of lactating women at 1, 3, 6, and 12 month of postpartum assessed by food frequency questionnaire
Concentration of human milk oligosaccharides, plant-based nutrients and fatty acids in breast milk | through study completion, an average of 1 year
  Breast milk composition by analyzing the concentration of human milk oligosaccharides, plant-based nutrients and fatty acids, using Liquid chromatography-mass spectrometry, Triple Quadrupole Mass Spectrometer, UV-Visible detector, flame ionization detector whichever appropriate, in the lactating women's breast milk collected at 3, 6, and 12 months postpartum.
Microbiota profiles | through study completion, an average of 1 year
  Microbiota profiles (microbiome operational taxonomic unit clustering and abundances, the Firmicutes/Bacteroidetes ratios, alpha and beta diversity) at 3, 6, and 12 month old by 16S ribosomal deoxyribonucleic acid sequencing

SECONDARY OUTCOMES:
Parameters of infant growth | through study completion, an average of 1 year
  The weight-for-age, length-for-age, BMI-for-age and head circumference-for-age, measured by a digital electronic balance, an infantometer and a measuring tape whichever appropriate, at 3, 6, and 12 month postpartum
Spherical-equivalent error and cylindrical error of infant | through study completion, an average of 1 year
  Refractive error of the infants at 6 and 12 month old measured in spherical-equivalent error and cylindrical error (diopter) by Autorefractor and Retinoscopy
Stereoacuity (sec of arc) of infant | through study completion, an average of 1 year
  Stereoacuity of the infants at 6 and 12 month old measured in stereoacuity (sec of arc) by Preschool Assessment of Stereopsis with a Smile test
Spatial frequency threshold of visual acuity of infant | through study completion, an average of 1 year
  Visual acuity (monocular and/or binocular) of the infants at 6 and 12 month old measured in spatial frequency threshold (cpd) by Lea Grating Paddles
Ocular deviation (prism diopter) of infant | through study completion, an average of 1 year
  Ocular alignment of the infants at 6 and 12 month old measured in Ocular deviation (prism diopter) by cover paddle and prism bar
The presence of secretor/lewis gene phenotypes of lactating women | through study completion, an average of 1 year
  At 3 month postpartum, mother's blood is collected. Genes that are related to breast milk oligosaccharide secretion including fucosyltransferase 2 and fucosyltransferase 3 will be accessed by polymerase chain reaction.
  The Secretor status and Lewis blood group of the mothers will be determined by the hemagglutination inhibition test. Hemagglutination will be examined using corresponding erythrocyte suspensions (3-5% erythrocytes in saline) and monoclonal anti-Lea and anti-Leb antibodies.
Untargeted metabolomics profiles of infant urine | through study completion, an average of 1 year
  Untargeted metabolomics profiling of infant urine at 3, 6, and 12 months old will be performed on an ultra-high performance liquid chromatography system coupled with high-resolution mass spectrometry.

CONTACTS AND LOCATIONS:
Overall Officials: Man Sau Wong, PhD, Principal Investigator — The Hong Kong Polytechnic University
Locations (1):
- The Hong Kong Polytechnic University, Hong Kong, China